CLINICAL TRIAL: NCT02057497
Title: An Exploratory Clinical Trial to Generate Whole Blood Samples for Analysing Genetic Polymorphisms Related to GPCR Dependent Signalling and the FTO Gene in Healthy Volunteers and in Patients With Diabetes
Brief Title: An Exploratory Clinical Trial to Generate Whole Blood Samples for Analysing Genetic Polymorphisms
Status: Withdrawn | Type: Observational
Why Stopped: It has been decided by the Sponsor not to conduct the trial.
Sponsor: Profil Institut für Stoffwechselforschung GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: OBDM-02
Record Dates: First submitted 2014-02-04; First posted 2014-02-07 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Prediabetes; Diabetes Type 1; Diabetes Type 2
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — whole blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Healthy volunteers: Considered generally healthy based on medical history and physical examination as per discretion of the investigator
- Type 1 Diabetes: T1DM diagnosed clinically prior to start of trial examinations
- Type 2 Diabetes: T2DM diagnosis prior to the start of trial examinations

SUMMARY:
G (guanine nucleotide binding) proteins associating with G protein-coupled receptors (GPCR) are key players in the pathogenesis of obesity and diabetes and are targets of pharmacotherapeutic inter-ventions. In addition, G proteins binding to GPCRs either directly or permissively determine the efficacy of lifestyle interventions and drugs aiming at weight management and diabetes treatment. Polymor-phisms of the fat mass and obesity-related protein (FTO) gene have been also well characterised and linked to energy intake, body fat mass as well as CVD risk and the susceptibility to weight-reducing interventions. Stratifying patients according to G protein and FTO-related genotyping may enable a more accurate prediction of individual disease courses and responses to therapeutic interventions in terms of safety and tolerability as well as efficacy. Although the objectives primarily refer to the analysis of G pro-tein and FTO-related genotypes, also other genes of potential relevance for the evolution of obesity and/ or diabetes and the response to lifestyle and pharmacological interventions may be analysed.

ELIGIBILITY:
Inclusion Criteria:

General

1. Informed consent obtained before any trial-related activities
2. Males and females equal or more than 18 years old Healthy volunteer-specific
3. Considered generally healthy based on medical history and physical examination as per discretion of the investigator

   T2DM-specific
4. T2DM diagnosis prior to the start of trial examinations.

   T1DM-specific
5. T1DM diagnosed clinically prior to start of trial examinations

Exclusion Criteria:

General

1. Mental incapacity or language barriers which preclude adequate understanding or cooperation, unwillingness to participate in the trial, known or suspected not to comply with trial directives or not to be reliable or trustworthy, or subjects who in the opinion of their general practitioner or the Investigator should not participate in the trial.

   Healthy volunteer-specific
2. Previous diagnosis of any type of diabetes mellitus, e.g. T1DM, T2DM, gestational diabetes, maturity onset diabetes of the young, etc.

   T2DM-specific
3. T1DM, diabetes resulting from pancreatic injury, or secondary forms of diabetes, e.g., acrome-galy or Cushing's syndrome.

   T1DM-specific
4. T2DM, diabetes resulting from pancreatic injury, or secondary forms of diabetes, e.g., acrome-galy or Cushing's syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers and patients with diabetes
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
Association of defined G protein- and FTO-related genotypes with the presence of T2DM or T1DM from a blood sample; also other genes of potential relevance for the evolution of obesity and/or diabetes. | day 1

SECONDARY OUTCOMES:
Association of defined G protein- and FTO-related genotypes with the T2DM risk of healthy volunteers from a blood sample. | day 1

CONTACTS AND LOCATIONS:
Overall Officials: Leona Plum-Mörschel, MD, Principal Investigator — Profil Institut fuer Stoffwechselforschung GmbH